CLINICAL TRIAL: NCT03811626
Title: Efficacy of Multidimensional Management of Mild Traumatic Brain Injury : A Randomised Clinical Trial
Brief Title: Efficacy of Multidimensional Management of Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche sur la Moelle épinière et l'Encéphale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012-A00015-38
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild TBI; quality of life; coping strategies; symptoms; neuropsychological tests; pain; memory reactive; Cognitive dimension
MeSH Terms: conditions — Brain Concussion; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patient who underwent cognitive-behavioral rehabilitation
  Interventions: Procedure: cognitive-behavioral rehabilitation
- Comparator (No Intervention): Patient with no specific management

INTERVENTIONS:
Procedure: cognitive-behavioral rehabilitation — Combination of clinical examination and neuropsychological and psychological tests
  Arms: Intervention

SUMMARY:
Unfavorable outcomes (UO) are seen in 15 to 20% of patients with mild traumatic brain injury (mTBI). Early identification of patients at risk for UO is crucial for suitable management to be initiated, increasing their chances for a return to a normal life. The investigators previously developed a diagnostic tool enabling early identification (8 to 21 days after the injury) of patients likely to develop UO. In the present study, the investigators examined the value and beneficial effects of early multidimensional management (MM) on prognosis. The investigators used a diagnostic tool to classify 221 mTBI patients as UO (97) or FO (favorable outcome) (124). Patients whose initial risk factors point to UO are at risk of developing post-concussion syndrome (PCS). UO patients were randomized into 2 groups: a group that underwent MM (cognitive-behavioral rehabilitation) (34) and a group with no specific management (46). At 6 months, these 2 groups were compared and the impact of MM on outcome was assessed. Among patients initially classified as FO (101), 95% had FO at 6 months and only 5 had PCS as defined by DSM-IV classification. Of the UO patients who received MM, 94% had no PCS 6 months after injury, whereas 52% of the UO patients who did not receive MM had persistent PCS. The effect of MM on the recovery of patients at 6 months, once adjusted for the main confounding factors, was statistically significant (p<0.001). These results show that the initiation of MM after early identification of at-risk mTBI patients can considerably improves their prognosis.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 18 to 65 who have suffered mTBI, have health care coverage, who understand French, who can be followed for 6 months, and who are able to understand, reply, and cooperate.

Exclusion Criteria:

* Patient intubated and/or ventilated and/or sedated upon arrival at hospital
* Patient with injury to the medulla and with neurological signs or multiple injuries (at least 1 of which is life-threatening)
* Brain injury incurred during a suicide attempt
* Patient presenting psychiatric or psychological disorders that are debilitating and/or interfere with follow-up and/or evaluation
* Psychoactive treatment ongoing at the time of injury
* History of hospitalization in specialized a psychiatric setting and/or sick leave for psychological reasons
* Patient with a neurological disorder
* Patient with substance dependence
* Subject under guardianship or wardship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | Baseline, 6 months -
  Change in quality of life assessed by QOLIBRI (Quality of Life after Brain Injury) Scale - QOLIBRI scale assess health-related quality of life (HRQoL) of individuals after traumatic brain injury. QOLIBRI is a comprehensive questionnaire with 37 items covering six dimensions of HRQoL after TBI. The QOLIBRI scores are reported on a 0-100 scale , where 0=worst possible quality of life and 100=best possible quality of life.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Chu Bicetre, Le Kremlin-Bicêtre
  - Chu Montpellier, Montpellier
  - Chu Bichat/Beaujon, Paris
  - CHU St ANTOINE, Paris
  - Chu Tenon, Paris
  - Chu Rouen, Rouen

REFERENCES:
- [Derived] Caplain S, Chenuc G, Blancho S, Marque S, Aghakhani N. Efficacy of Psychoeducation and Cognitive Rehabilitation After Mild Traumatic Brain Injury for Preventing Post-concussional Syndrome in Individuals With High Risk of Poor Prognosis: A Randomized Clinical Trial. Front Neurol. 2019 Sep 4;10:929. doi: 10.3389/fneur.2019.00929. eCollection 2019. PMID 31551902
- See also: Early Detection of Poor Outcome after Mild Traumatic Brain Injury: Predictive Factors Using a Multidimensional Approach a Pilot Study. — https://www.ncbi.nlm.nih.gov/pubmed/29312112